CLINICAL TRIAL: NCT06933849
Title: PartnerED Care: Coordinated Emergency Department Transitions for Assisted Living Patients With Alzheimer's Disease and Related Dementias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ellen McCreedy, Associate Professor, Brown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U54AG063546_Pilot Cycle 5A; U54AG063546 (NIH)
Record Dates: First submitted 2025-03-30; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease or Associated Disorder
Keywords: case management; emergency department; feasibility
MeSH Terms: conditions — Alzheimer Disease; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients with eligible emergency department visits between November 1, 2023 and June 30, 2024 (Experimental)
  Interventions: Behavioral: Structured case management

INTERVENTIONS:
Behavioral: Structured case management — When a Bluestone Accountable Care Organization registers in an emergency department, a Bluestone chronic care manager contacts emergency department clinicians by phone and fax to provide up-to-date clinical and discharge support information.

SUMMARY:
The goal of this observational study is to learn the feasibility, acceptability, appropriateness, and adherence to a case management intervention. PartnerED is a case management intervention that aims to reduce unnecessary hospital admissions by providing real-time, structured information and discharge support to emergency department providers via phone and fax. The intervention is led by chronic care managers employed by Bluestone Accountable Care Organization, a physician group primarily serving patients in assisted living centers.

ELIGIBILITY:
Inclusion Criteria:

* Bluestone Accountable Care Organization patient
* Registration in emergency department between November 1, 2023 and June 30, 2024, as recorded in electronic admission, discharge, and transfer notifications

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1989 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Percent of eligible emergency department visits with completed outreach | Within 1-3 hours of emergency department registration
  Percent of eligible emergency department visits in which a case manager provided structured clinical and discharge support information to a emergency department provider about a patient who was in their care, with the goal of avoiding an unnecessary hospitalization

SECONDARY OUTCOMES:
Percent of successful outreach conversations in which staff reported avoidance of an unnecessary hospitalization | Within 24 hours of emergency department registration
  Case manager self-report of whether she/he was successful in avoiding an unnecessary hospitalization of a patient after providing structured clinical and discharge support information to the emergency department provider

CONTACTS AND LOCATIONS:
Overall Officials: Ellen McCreedy, PhD, MPH, Principal Investigator — Brown University
Locations (1):
- Bluestone Accountable Care Organization, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Data use agreements do not allow for sharing individual participant data